CLINICAL TRIAL: NCT00902434
Title: Retrospective Analysis of Histologies, Pattern of Care, and Outcomes of Non-Hodgkin Lymphoma in Elderly Patients Above the Age of 80 in the Rituximab Era: A Report From the Chicago Lymphoma Consortium
Brief Title: Non-Hodgkin Lymphoma in Elderly Patients Above the Age of 80 in the Rituximab Era
Status: Completed | Type: Observational
Sponsor: Oncology Specialists, S.C. (Other)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Other Study IDs: 0903
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an exploratory analysis that is investigating the pattern of care in patients over the age of 80 who were diagnosed with non-Hodgkin lymphoma (NHL). This study will look at the dose intensity and density implemented in this patient population to calculate whether patients received the full course of therapy, received less duration of treatment, or received lower doses of the drugs administered. Furthermore, the investigators would explore time to disease progression for these patients regardless of the treatment received and investigate whether patient outcomes differ based on the type of therapy or dose intensity/density given.

This study is looking at retrospectively evaluating patients with NHL who are over the age of 80 at our institution between 2001-2007. It is anticipated that about 50 patients will be included in this study.

DETAILED DESCRIPTION:
Non-Hodgkin Lymphoma (NHL) is a malignant disease of the lymphoid and hematopoetic system with an annual incidence of 60,000 cases/year in the United States accounting for over 18,000 deaths annually. NHL is a heterogeneous malignancy with a median age of 65 at the time of diagnosis. Most clinical trials that have established current standards of care did not include elderly patients, especially those who are above the age of 80. Reasons for such under representation are not well-defined but several factors are hypothesized. Patients above the age of 80 have many co-morbid conditions that might exclude them from enrollment on clinical studies that are usually designed for more fit individuals. In addition, investigators are often reluctant to propose trials to elderly patients as their response to therapy might be suboptimal compared with younger patients affecting the overall data.

Well-designed published studies as to how patients over the age of 80 are being managed in the community or academic setting are lacking. There is no agreed-upon treatment algorithm for these patients and recommended approach varies based on the treating physician, the institution, and each individual patient.

Some physicians chose to offer dose reductions while others might omit chemotherapy and use monoclonal antibodies alone. Furthermore, treatment duration and the number of cycles given might vary considerably in this patient subgroup for a variety of reasons, mainly toxicity. In addition, it is unclear whether the histologic distribution of NHL is similar in older patients. In other words, it is not clear whether patients over the age of 80 are commonly diagnosed with diffuse large cell lymphoma (DLCL) and follicular lymphoma (FL) similar to younger individuals. Most importantly, these expected variations in treatment strategies might have inferior outcomes when compared to younger patient population. Looking at histologic subtype, treatment strategies, and outcomes in patients over the age of 80 is useful for patients and physicians alike. It is plausible that our current standards do not apply to this very-older patient population arguing for offering them clinical trials or novel agents even as an initial approach. On the other hand, we might discover that these older patients fare well despite these variations arguing that their disease biology is different especially if we note changes in histologic distribution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any NHL diagnosis regardless of histology who are over the age of 80 at the time of diagnosis will be included and analyzed.
* Data on age, gender, performance status, and major co-morbid conditions will be collected.
* Histology of the diagnosed NHL will be recorded. The grade (1, 2, or 3) for those who were diagnosed with follicular lymphoma will also be recorded.
* Stage of the disease, presence of bulky nodes and B symptoms will also be recorded.
* PET scan results if available.
* Type of treatment received will be recorded.
* Responses to therapy.
* Outcomes of treatment implemented and toxicities incurred.
* Subsequent therapies if applicable.

Exclusion Criteria:

* None. All charts of patients who are above the age of 80 at the time of NHL diagnosis will be analyzed.

Ages: 80 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study is looking at retrospectively evaluating patients with NHL who are over the age of 80 at our institution between 2001-2007.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, S.C.